CLINICAL TRIAL: NCT04958200
Title: Integrated Technology-Based Intervention to Reduce Heavy Drinking and Chronic Pain Among Patients in Primary Care
Brief Title: Alcohol Use and Chronic Pain Among Primary Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Tibor Palfai, Professor of Psychological and Brain Sciences, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4947; R34AA027598-01 (NIH)
Record Dates: First submitted 2021-06-30; First posted 2021-07-12 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Alcohol Drinking; Chronic Pain
MeSH Terms: conditions — Alcohol Drinking; Chronic Pain | interventions — Ethanol; Therapeutics

STUDY DESIGN:
Intervention Model Description: Compare intervention to a treatment as usual comparison condition
Who Masked: Outcomes Assessor
Masking Description: Eight-week and 16-week assessments will be completed by assessor who is masked to intervention condition. Baseline assessment takes place before randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mhealth-pc for alcohol and chronic pain (Experimental): Smartphone-based intervention
  Interventions: Behavioral: mhealth-pc for alcohol and pain
- Treatment As Usual (Active Comparator): In person session that provides enhanced treatment as usual
  Interventions: Behavioral: Treatment As Usual

INTERVENTIONS:
Behavioral: mhealth-pc for alcohol and pain — Smartphone-based intervention that includes in-person initial session and 8 video lessons, daily activities, and weekly check-ins.
  Arms: mhealth-pc for alcohol and chronic pain
Behavioral: Treatment As Usual — psychoeducation on pain and alcohol use and treatment resource information
  Arms: Treatment As Usual

SUMMARY:
Chronic pain and unhealthy drinking are common co-occurring conditions among patients presenting to primary care. Given their impact on functioning and medical outcomes, there would be considerable benefit to developing an accessible, easily utilized, integrative approach to reduce unhealthy alcohol use and pain that can be readily incorporated into the primary care setting. The objective of this study is to test a smartphone-based intervention for reducing unhealthy alcohol use and pain in primary care patients, determine the feasibility of implementing this intervention in the primary care setting, provide effect size estimates of the intervention on drinking and chronic pain outcomes.

DETAILED DESCRIPTION:
Heavy alcohol use represents a significant risk for morbidity and mortality. Unfortunately, addressing unhealthy patterns of alcohol use in primary care is often a challenge as patients typically present with co-morbid conditions that: (1) may make unhealthy drinking a lower priority health issue and (2) may impact the capacity for sustained alcohol-related change. Chronic pain is among the most common of these conditions among primary care patients. Pain is a frequent source of distress and disability among primary care patients and is one of the most frequent causes for visits. Pain is also an important trigger for alcohol use among primary care patients who drink and is associated with the experience of negative alcohol-related consequences and unhealthy drinking over time. The experience of pain has also been shown to be associated with poorer responses to alcohol interventions. Primary care physicians face a number of challenges when attempting to treat co-occurring unhealthy drinking and pain among their patients. Pain management and reduction of alcohol use among those who engage in heavy alcohol use is often not adequately achieved with pharmacological treatments nor are pharmacological treatments indicated for common pain conditions. Moreover, despite the availability of evidence-based psychosocial interventions for unhealthy drinking and chronic pain, patients with each of these conditions typically show poor adherence to treatment. Given the rates of pain and unhealthy alcohol use among primary care patients and their impact on functioning and medical outcomes, there would be considerable benefit to an accessible, easily utilized, integrative approach to treat heavy alcohol use and pain that can be readily incorporated into the primary care setting. The objectives of this study are to develop a smartphone-based intervention for reducing heavy alcohol use and pain in primary care patients, determine the feasibility of implementing this intervention in the primary care setting, provide effect size estimates of the intervention on outcomes, and develop procedures to conduct a Stage II efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

* 1 heavy drinking: defined as either [1] an average of more than 7(for women)/14 (for men) standard drinks per week over the past month or [2] one or more heavy drinking episodes (4+ standard drinks for women, 5+ standard drinks for men)
* 2 chronic pain: defined as non-cancer related pain of at least 3 months duration rated as moderate or greater (past week pain severity rating of 4 or greater on the BPI severity item)

Exclusion Criteria:

* psychoactive medication for pain or alcohol use for fewer than 2 months
* history of bipolar disorder or schizophenia
* current expressed suicidal intent
* prior history of alcohol withdrawal related seizures or delirium tremens
* behavioral treatment for pain or alcohol use in the past 3 months
* any scheduled surgery within the next 6 months or acute life threatening illness that requires treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Boston University Department of Psychological and Brain Sciences, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing procedures that will be implemented within one year of completion of the study. Specific data may be shared based on proposals received and reviewed by the study investigators and limited public-use data sets might be prepared and made available. In either case, data will be shared only after all planned reports of study findings have been prepared. Data to be shared will be de-identified to minimize the risk of deductive disclosure. Documentation will be provided for all shared data including copies of data collection forms, schedule of study assessments, data dictionaries documenting all original and derived variables, descriptive statistics for all variables included in the data sets, and a written description of the study conduct and noteworthy details anticipated to potentially affect data interpretation. Costs associated with producing data sets and analysis will be the responsibility of investigators seeking the data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after all planned reports of study findings have been prepared within one year of project completion. Data will be available upon request for 5 years following these reports
Access Criteria: Specific data may be shared based on proposals received and reviewed by the study investigators and determined to have scientific merit.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 49 participants who signed to consent form. One person decided NOT to participate post-consent and therefore did not complete any baseline information or get randomized to condition. Therefore only 48 completed baseline and were randomized to condition
Period: Overall Study
Arm/Group | Mhealth-pc for Alcohol and Chronic Pain | Treatment As Usual
Started | 24 | 24
Completed | 21 | 20
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Population: A total of 49 participants signed the study consent form. One participant withdrew post consent, prior to baseline assessment and randomization to condition. Consequently, there were baseline data collected for only 48 participants who were all randomized to condition
Groups:
- Total: Total of all reporting groups
Arm/Group | Mhealth-pc for Alcohol and Chronic Pain | Treatment As Usual | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 18 | 37
  >=65 years | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.17 (13.15) | 52.42 (17.35) | 52.79 (15.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 10 | 10 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 20 | 20 | 40
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 48
Number of heavy drinking episode days in the past 30 days [Mean (Standard Deviation); unit: heavy drinking days] | 11.25 (11.78) | 8.79 (8.93) | 10.02 (10.41)
Average number of drinks per week over the past 30 days [Mean (Standard Deviation); unit: drinks/week] | 22.33 (22.27) | 18.36 (15.89) | 20.35 (19.24)
Pain, Enjoyment, General Activity (PEG) [Mean (Standard Deviation); unit: units on a scale] — This scale consists of 3-items that range from 0-10 each. The overall pain score on the PEG is the mean of these 3 items. The possible range is 0-10 with higher scores reflecting a worse outcome (i.e., more pain).
  units on a scale | 6.36 (1.69) | 5.76 (1.83) | 6.06 (1.77)
Pain Intensity: Brief Pain Inventory [Mean (Standard Deviation); unit: units on a scale] — This scale consists of 4-items that range from 0-10 each. The overall pain score on the pain severity score is the mean of these 4 items. The possible range is 0-10 with higher scores reflecting a worse outcome (i.e., more severe pain).
  units on a scale | 5.4 (1.71) | 4.66 (1.46) | 5.03 (1.61)
Pain Interference: Brief Pain Inventory [Mean (Standard Deviation); unit: units on a scale] — This scale consists of 7-items that range from 0-10 each. The overall pain interference score is the mean of these 7 items. The possible range is 0-10 with higher scores reflecting a worse outcome (i.e., more pain interference).
  units on a scale | 6.21 (1.88) | 5.24 (2.15) | 5.72 (2.06)

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Time Line Followback (30)- Heavy Drinking Episode Days in the Past 30 Days
Description: Number of heavy drinking episode days (i.e., days with consumption of 5+ drinks men/4+ drinks women)
Time Frame: Past 30 days as assessed at the 16-week timepoint
Population: multiple imputation was used in analyses for primary outcomes only
Measure: Mean (Standard Deviation); unit: heavy drinking days
Arm/Group | Mhealth-pc for Alcohol and Chronic Pain | Treatment As Usual
Number analyzed (Participants) | 24 | 24
heavy drinking days | 7.9 (11.32) | 4.3 (5.57)

2. Primary Outcome: Alcohol Time Line Followback (30)- Average Drinks Per Week in the Past 30 Days
Description: Average number of standard alcohol-containing drinks per week over the past 30 days
Time Frame: Past 30 days as assessed at the 16-week timepoint
Measure: Mean (Standard Deviation); unit: drinks per week
Arm/Group | Mhealth-pc for Alcohol and Chronic Pain | Treatment As Usual
Number analyzed (Participants) | 24 | 24
drinks per week | 16.89 (20.60) | 10.56 (9.02)

3. Primary Outcome: The Pain, Enjoyment of Life, General Activity (PEG) Scale
Description: Three items which assess chronic pain intensity and interference. Range of each item is 0-10. Mean rating of the three items indicate the PEG pain score. range of scale is 0-10. Higher scores reflect worse outcomes
Time Frame: Past 7 days as assessed at the 16-week timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mhealth-pc for Alcohol and Chronic Pain | Treatment As Usual
Number analyzed (Participants) | 24 | 24
score on a scale | 4.60 (2.56) | 4.82 (1.79)

4. Secondary Outcome: Pain Intensity - Brief Pain Inventory (BPI) Items
Description: Four items from the Brief Pain Inventory (BPI) comprise the pain severity subscale. Pain severity score reflects the mean item rating of these 4 items. Range 0-10.
  Higher scores reflect worse outcomes.
Time Frame: past 7 days as assessed at the 16-week timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mhealth-pc for Alcohol and Chronic Pain | Treatment As Usual
Number analyzed (Participants) | 21 | 20
score on a scale | 3.98 (1.93) | 4.16 (1.21)

5. Secondary Outcome: Pain Interference
Description: Seven items from the BPI are used to assess chronic pain interference. Each item is 0-10. The pain interference score is the mean of these seven items and ranges from 0-10.
  Higher scores reflect worse outcomes
Time Frame: past 7 days as assessed at the 16-week timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mhealth-pc for Alcohol and Chronic Pain | Treatment As Usual
Number analyzed (Participants) | 21 | 20
score on a scale | 4.37 (2.63) | 4.68 (2.36)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the period in which the participant was in the study which was 16-weeks.
Arm/Group | Mhealth-pc for Alcohol and Chronic Pain | Treatment As Usual
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 1/24
Other Adverse Events (participants affected / at risk) | 1/24 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mhealth-pc for Alcohol and Chronic Pain (N=24) | Treatment As Usual (N=24)
Hospitalization (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — participant hospitalized for car accident....broken bones in feet...not study related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mhealth-pc for Alcohol and Chronic Pain (N=24) | Treatment As Usual (N=24)
hospital visit for uncontrolled diabetes (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — diabetes regulated after visit to hospital

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT04958200/Prot_SAP_000.pdf
  • Informed Consent Form (2024-09-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT04958200/ICF_001.pdf